CLINICAL TRIAL: NCT04747041
Title: Evaluation of a Phyto Aromatherapy Treatment in the Management of Recurrent Cystitis Preliminary Study
Brief Title: Evaluation of a Phyto Aromatherapy Treatment in the Management of Recurrent Cystitis
Acronym: CYSTALTERNA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-AOIP-02
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cystitis Recurrent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alternating each month for 1 year between Phytocyst herbal tea and Cyscontrol (Experimental): Alternating each month (From Day1 to DAY15) for 1 year between Phytocyst herbal tea and Cyscontrol = Preventive Treatment In case of episode of cystitis : AROMAFEMINA, Capsules for the comfort of the urinary tract Oleocaps 2 : 2 capsules before meals, 3 times a day for 5 consecutive days.
  Interventions: Combination Product: CYSCONTROL/PHYTOCYST Herbal tea

INTERVENTIONS:
Combination Product: CYSCONTROL/PHYTOCYST Herbal tea — Alternating every month from Day1 to Day15 cyscontrol and phytocyst herbal tea to prevent episode of cystitis

SUMMARY:
Half of the women have a once-in-a-lifetime episode of cystitis. Recurrence occurs in about 20% to 30% of patients, and half of these patients will have more than 4 episodes per year, defining recurrent cystitis.

The clinical assessment sometimes brings to light favourable factors; variables in pre- or post-menopause; but in the majority of cases, no explanatory cause can solve the problem and some authors refer to resignation as a classic reaction to this problem.

several countries have already opted for alternative treatments (Nonsteroidal anti-inflammatory drugs, phytotherapy, diuresis treatment), especially since the pressure of antibiotic selection is at the root of the dramatic spread of bacterial resistances.

There is a growing interest in the potential of complementary medicine to assist in this care. Products based on cranberries, for example, have been particularly studied and a 2012 Cochrane review concluded that there is a benefit with an estimated risk reduction of between 10 and 20%. Another "alternative" approach is the use of Chinese medicinal herbs. These herbs have been used for more than 2000 years.

The implementation of phyto-aromatherapy treatment implies a global management of patients with recurrent cystitis. Initially, it involves a curative phase as soon as the first symptoms of the attack appear, thanks to a mixture of antibacterial essential oils. In a second phase, it integrates a preventive phase over several months thanks to an association of medicinal plants whose effects in this field have been proven in vitro and in vivo, allowing to rebalance a "terrain" associating anxiety, hypersensitivity to pain, a terrain willingly associated with the irritable bowel syndrome in these patients. While having few side effects, the plants will act, in the long term, at different levels: directly on the cause of the disease thanks to their antiseptic, antiadhesive and diuretic activities, but also by reducing the symptoms thanks to their anti-inflammatory, analgesic, antispasmodic and anxiolytic activities.

Investigators hypothesize that patients with recurrent cystitis can be improved by a two-phase, multi-plant, phyto-aromatherapy treatment combining several plants: the treatment of attacks, by aromatherapy, and a prophylactic treatment, by phytotherapy. In the absence of any such studies published in the literature, investigators propose a non-randomised prospective monocentric interventional pilot study on 15 patients with proof of concept and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older.
* Affiliated to social security.
* Presenting recurrent cystitis defined by a frequency of at least 4 episodes per year.
* For women of childbearing age: effective contraception followed for at least 3 months prior to the start of the study and agreeing to keep it throughout the study period
* Available to consult a phyto-aromatherapy pharmacist for an initial consultation and then every 3 months (M3, 6,9, 12) and then at 18 months.
* Having been previously explored according to good practice and informed
* Having signed the informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Severe visceral deficiencies in the previous year.
* Individualised psychiatric pathology.
* Other progressive infectious pathologies requiring antibiotic treatment.
* Taking anticoagulants.
* Concomitant intake of non-drug treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
adherence to phyto-aromatherapy treatment | 12th month
  The scale called "treatment compliance" ranges from 1 to 10. A score of 1 means not at all observant and 10 means very observant.

SECONDARY OUTCOMES:
Antibiotic treatments | 12 months
  The number of antibiotic treatments over 12 months
Number of cystitis | 12 months
  The number of cystitis over the 12 months of the protocol
Patients' overall satisfaction | 12 months
  Patients' overall satisfaction will be assessed on a simple numerical scale from 1 to 10. The scale is called the "General Satisfaction Scale" and ranges from 1 to 10. A score of 1 means not at all satisfied and 10 means very satisfied. As well as their ability to manage their symptoms. Three analogue scales will also be used to assess the impact of the protocol on patients' sexuality (including anxiety and comfort in relation to intercourse, when appropriate)
Recording adverse events | 18 months
  The nature of the side effects, sought and at each phyto-aromatherapy consultation
The benefit persisting at 6 months after stopping treatment with phyto-aromatherapy | During 6 months after stopping treatment (patient stop treatment at Month12 so between the 12th and 18th month)
  The benefit persisting at 6 months after stopping treatment with phyto-aromatherapy will be evaluated on the number of times antibiotic therapy is used over a period of 6 months after stopping the treatment
Evaluation of the evolution of bacterial resistance on phenotypes isolated from the cytobacteriological examination of urine | From date of inclusion until the date of documented episode of cystitis, assessed up to 18 months
  Evaluation of the evolution of bacterial resistance on phenotypes isolated from the cytobacteriological examination of urine if inclusion resistance markers are present, in comparison with the last cytobacteriological examination of urine carried out during the protocol period, requested in the event of a clinical episode. A cytobacteriological examination of the urine carried out on a systematic basis that can detect asymptomatic colonisation or bacteriuria is not appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique MONDAIN, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Archet, Nice, France